CLINICAL TRIAL: NCT04116827
Title: Analysis of Sleep and Activity Patterns in Pre-menopausal Breast Cancer Patients After Taking Tamoxifen Using a Wrist-worn Internet of Things Device
Brief Title: Sleep and Activity Patterns in Pre-menopausal Breast Cancer Patients on Tamoxifen Using a Wrist-worn Internet of Things Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor of Physical and Rehabilitation Medicine, Samsung Medical Center
Other Study IDs: SMC 2018-07-014-011
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Sleep Disorder; Breast Cancer
Keywords: sleep disorder; breast cancer; pre-menopausal; tamoxifen; hormone therapy
MeSH Terms: conditions — Sleep Wake Disorders; Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tamoxifen group: Pre-menopausal breast cancer patients who underwent proper surgical treatment, chemotherapy, or radiation therapy, and are scheduled for application of tamoxifen and goserelin
  Interventions: Drug: Tamoxifen Oral Tablet

INTERVENTIONS:
Drug: Tamoxifen Oral Tablet — Patients who are scheduled for application of tamoxifen and goserelin

SUMMARY:
The aim of this study is to observe the sleep and activity patterns of pre-menopausal breast cancer patients taking tamoxifen using a wrist-worn internet of things device and questionnaires.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumors occurring in women worldwide. Treatments include surgery, radiation therapy, chemotherapy, hormone therapy, and target therapy. As multidisciplinary treatment improves breast cancer survival, there is a growing interest in the quality of life of breast cancer survivors. Common symptoms that patients with breast cancer continue to complain of during or after their treatment include fatigue, pain, depression, sleep disorders, weight gain and hot flashes.

There are only a few studies investigating sleep problems in breast cancer patients, which mostly relied on surveys. A commonly used survey evaluation method is the Pittsburg Sleep Quality Index (PSQI). Using PSQI, one study reported that 66% of the Chinese breast cancer survivors had sleep disorders and 49% had significantly reduced sleep efficiency and time in bed. The group with sleep disorder had lower quality of life, more depression and higher overall stress than the group without sleep disorder. Another survey of breast cancer patients over 69 years old found that pain, fatigue and depression were related to sleep, and that fatigue was the strongest predictor of sleep disorders.

A recent study found that postmenopausal breast cancer patients, starting hormone therapy with aromatase inhibitor, total sleep time and sleep efficiency declined without statistical significance. However, 58% of Korean breast cancer patients are pre-menopausal patients aged 49 or younger, and thus, most patients take tamoxifen and goserelin instead of aromatase inhibitors after surgery. In this reason, results of aromatase inhibitor can not be applied in this population. As previous studies on the effects of tamoxifen on sleep were conducted retrospectively, objective comparisons of before and after applying tamoxifen are difficult and the long-term effects of tamoxifen are difficult to understand.

The aim of this study is to observe the sleep and activity patterns of pre-menopausal breast cancer patients taking tamoxifen using a wrist-worn internet of things device and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of unilateral breast cancer (stage 0 ~III)
* underwent proper cancer treatment including surgery, chemotherapy, radiation therapy
* age : 18 ~ 45
* scheduled for applying tamoxifen and goserelin

Exclusion Criteria:

* need CPAP device during sleep due to sleep apnea
* under medication for restless leg syndrome
* previous history of tamoxifen
* irregular bedtime due to shift work
* diagnosed of recurrent or metastatic cancer
* have difficulty understanding and conducting surveys and verbal instructions due to severe cognitive, communication and perception problems
* refuse to participate
* has musculoskeletal system and neurological damage and lesions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female population, aged 18~45, diagnosed of unilateral breast cancer (stage 0 ~III), who underwent proper cancer treatment including surgery, chemotherapy, radiation therapy, scheduled for applying tamoxifen and goserelin
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
total sleep time | study enroll~12 months
  mean total sleep time per day, recorded by wrist-worn IoT device
walking steps and walking time | study enroll~12 months
  mean walking steps and walking time per day, recorded by wrist-worn IoT device

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | study enroll~12 months
  questionnaire developed to evaluate quality of sleep and sleep disorder
Insomnia Severity Index (ISI) | study enroll~12 months
  questionnaire developed to evaluate insomnia
Distress thermometer | study enroll~12 months
  well-known screening tool for psycho-social distress of cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azim HA Jr, Davidson NE, Ruddy KJ. Challenges in Treating Premenopausal Women with Endocrine-Sensitive Breast Cancer. Am Soc Clin Oncol Educ Book. 2016;35:23-32. doi: 10.1200/EDBK_159069. PMID 27249683
- [Background] Gonzalez BD, Lu Q. Sleep disturbance among Chinese breast cancer survivors living in the USA. Support Care Cancer. 2018 Jun;26(6):1695-1698. doi: 10.1007/s00520-018-4128-y. Epub 2018 Feb 26. PMID 29484499
- [Result] Bhave MA, Speth KA, Kidwell KM, Lyden A, Alsamarraie C, Murphy SL, Henry NL. Effect of Aromatase Inhibitor Therapy on Sleep and Activity Patterns in Early-stage Breast Cancer. Clin Breast Cancer. 2018 Apr;18(2):168-174.e2. doi: 10.1016/j.clbc.2017.12.012. Epub 2017 Dec 27. PMID 29361424
- [Result] Budhrani PH, Lengacher CA, Kip K, Tofthagen C, Jim H. An integrative review of subjective and objective measures of sleep disturbances in breast cancer survivors. Clin J Oncol Nurs. 2015 Apr;19(2):185-91. doi: 10.1188/15.CJON.185-191. PMID 25840384
- [Result] Chen D, Yin Z, Fang B. Measurements and status of sleep quality in patients with cancers. Support Care Cancer. 2018 Feb;26(2):405-414. doi: 10.1007/s00520-017-3927-x. Epub 2017 Oct 23. PMID 29058128
- [Result] Yfantis A, Intas G, Tolia M, Nikolaou M, Tsoukalas N, Lymperi M, Kyrgias G, Zografos G, Kontos M. Health-related quality of life of young women with breast cancer. Review of the literature. J BUON. 2018 Jan-Feb;23(1):1-6. PMID 29552751
- [Derived] Yeo SM, Lim JY, Kim SW, Chae BJ, Yu J, Ryu JM, Hwang JH. Impact of Adjuvant Hormone Therapy on Sleep, Physical Activity, and Quality of Life in Premenopausal Breast Cancer: 12-Month Observational Study. J Breast Cancer. 2023 Apr;26(2):93-104. doi: 10.4048/jbc.2023.26.e11. Epub 2023 Mar 13. PMID 37051646